CLINICAL TRIAL: NCT05272592
Title: Protocol for CAMUS Nurse Delphi Study: Active Involvement of Nursing Staff in Reporting and Grading Complication-Intervention Events - An Approach to Improve Patient Safety and Quality of Surgical Care
Brief Title: Protocol for CAMUS Nurse Delphi Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2022.046
Record Dates: First submitted 2022-02-18; First posted 2022-03-09 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Perioperative/Postoperative Complications; Urologic Diseases
MeSH Terms: conditions — Postoperative Complications; Urologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing staff: Certified local-and-international inpatient-and-outpatient nurses specialised in urology, perioperative nurses, and urology-specific advanced practice nurses/nurse practitioners will be included.

SUMMARY:
Multi-staged, international Nurse Delphi study that aims to validate the newly proposed CAMUS System and CAMUS CCI in an experienced nursing staff population.

DETAILED DESCRIPTION:
Background: Comprehensive and reproducible assessment of post-operative complications are essential for reliable evaluation of quality of care and subsequent reformation of hospital safety infrastructure. At present, significant discrepancies exist in complication reporting and grading, and current complication systems lack holistic assessment of patient care by failing to consider and incorporate nursing insight and perception of patient burden.

Objective: To gain experienced nursing perspective on current and future complication reporting and grading in Urology, validate the CAMUS-CCI, and quality control the use of the CDC in nurses.

Design, Setting, and Participants: The 12 part REDCap-based Delphi survey was developed in conjunction with methodologist review, experienced nursing and urologist opinion. Certified local and international inpatient and outpatient nurses specialised in urology, perioperative nurses, and urology-specific advanced practice nurses/nurse practitioners will be included. A minimum sample size of 250 participants is targeted.

Outcome Measurements and Statistical Analysis: The survey assesses participant demographics, nursing experience and opinion on complication reporting and the proposed CAMUS reporting recommendations, grading of intervention events using the existing Clavien-Dindo Classification and the proposed CAMUS Classification, and rating various clinical scenarios. Consensus will be defined as ≥75% agreement. If consensus is not reached, subsequent Delphi rounds will be performed under Steering Committee guidance.

ELIGIBILITY:
Inclusion Criteria:

* Certified nurses
* Local or international nurses
* Inpatient or outpatient nurses
* Peri-operative nurses
* Urology-specific advanced practice nurses/nurse practitioners

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Certified local-and-international inpatient-and-outpatient nurses specialised in urology, perioperative nurses, and urology-specific advanced practice nurses/nurse practitioners will be included.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Validation of the newly proposed CAMUS System and CAMUS CCI in an experienced nursing staff population | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Furrer, MD, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided